CLINICAL TRIAL: NCT02252666
Title: Exploring the Use of Non-invasive Neuromodulation Combined With Exercise in People With Advanced Multiple Sclerosis (MS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-1060
Record Dates: First submitted 2014-07-15; First posted 2014-09-30 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Multiple Sclerosis
Keywords: MS; balance; standing; control; movement
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Neuromodulation Rehabilitation (Experimental): Balance, posture and gait activities; therapeutic exercise for isolated muscle control; transfer training; and relaxation training using neurostimulation modulation. 2-week in lab intervention training, training at home and periodic return for follow-up testing and instruction on the next phase of the intervention.
  Interventions: Device: Neuromodulation Rehabilitation

INTERVENTIONS:
Device: Neuromodulation Rehabilitation — CN-NINM uses sequenced patterns of electrical stimulation on the tongue. Our hypothesis is that CN-NINM induces neuroplasticity by noninvasive stimulation of two major cranial nerves: trigeminal, CN-V, and facial, CN-VII.
  Other Names: Cranial Nerve Non-invasive Neuromodulation (CN-NINM); Portable Neuromodulation Stimulator (PoNS)

SUMMARY:
The investigators hypothesis is that electrical stimulation to the tongue that directly stimulates two cranial nerve nuclei (Trigeminal and Facial Nerve Nuclei), will excite neural impulses to the brainstem and cerebellum. The investigators call this cranial nerve non-invasive neuromodulation (CN-NINM). The activation of these structures induces neuroplasticity when combined with specific physical exercises, can reduce symptoms of advanced MS, targeting primarily postural stability (sitting and standing), upper extremity movement, and ability to perform self-transfers.

DETAILED DESCRIPTION:
The intervention will be similar to that used in the investigators previous work with movement disorders, and will be tailored to the address issues unique to individuals with advanced MS.

The study will enroll a total of 6 subjects having advanced MS that present with significant seated and standing balance, posture, or movement control deficits due to MS.

Subjects will complete twice-daily lab training for two weeks (5 days/week). Each lab training (morning and afternoon) includes 1.5 to 2 hours of instruction in balance, posture and gait activities; therapeutic exercise for isolated muscle control; transfer training; and relaxation training.

Activities are performed in 20-minute sessions with concomitant electrical stimulation of the tongue. The intervention is customized according to each subject's particular symptoms and tolerance. If a subject is not able to perform this amount of training, the training will be adapted to a level that is tolerable.

After these 2 weeks, subjects will continue to perform these same intervention activities at home for 4 weeks. They will return to the lab for 1 week of training and testing, then perform home training for 4 weeks. This cycle is repeated for a total of 5 cycles.

After the 6 months have been completed, subjects may choose to participate in an optional second phase of the study. The second phase includes an additional 12 months of participation in which subjects perform the intervention activities at home training and return to the lab on time per month for 2 hours of testing and 2 hours of training.

If successful, this study would indicate that CN-NINM intervention may reduce the symptoms of advanced MS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be age 18 or older.
* Subjects will have a score between 6.5 to 7.5 on the Kurtzke Expanded Disability Status Scale (EDSS). The EDSS is a method of quantifying disability in people with multiple sclerosis.

  * Score of 6.5: needs constant bilateral support to walk 20 meters without resting.
  * Score of 7.0: unable to walk beyond five meters even with aid, and is essentially restricted to a wheelchair; wheels self and transfers alone, and is active in wheelchair about 12 hours a day.
  * Score of 7.5: unable to take more than a few steps and is restricted to wheelchair, and may need aid to transfer; wheels self, but may require a motorized chair for a full day's activities.
* Subjects will have reached a plateau in an MS focused physical rehabilitation program in the 6 months prior to enrollment.

  * Requiring prior physical therapy will ensure that subjects have a core level of function that will allow them to participate in the study.
  * Requiring that subjects have reached a plateau will ensure that subjects' response to the intervention is due to the use of the device and not to the physical exercises alone.
  * Subjects who have participated in a physical rehabilitation program demonstrate that they are willing and able to commit to a rigorous training regimen.
* Subjects will have a maximum score of 20 on the Trunk Impairment Scale (TIS). The TIS assesses static dynamic sitting balance and trunk coordination in a sitting position. A score of 20 or lower indicates that their ability to adequately maintain sitting posture is affected.
* Subjects may have upper extremity involvement.
* Subjects may have additional symptoms of nystagmus, dysarthria, sensory disturbance, pain, and/or bowel and bladder function. As they present, we will use appropriate assessments at baseline and successive study test points.
* Subjects are their own legal guardians, and are able to understand and give informed consent.

Exclusion Criteria:

Subjects will have no major co-morbidities, especially neurological disorders, uncontrolled pain, hypertension or diabetes. All subjects, if on medications, will not have had any major changes in type or dosage in within 3 months of enrollment. Additionally, candidates will be excluded if they:

* have Functional Systems Scores (FSS) 4 or greater for pyramidal, cerebellar, brainstem, and sensory functions; 3 or greater for bowel and bladder function; and 2 or greater for cerebral function;
* are able to walk independently;
* use tobacco products (these activities tend to reduce tactile sensitivity in the oral cavity);
* have any oral abrasions, cuts, cold sores, piercings, tissue inflammation, or have had oral surgery within the previous 3 months;
* have a pacemaker, or are identified as at-risk for cardiovascular events;
* have a history of seizures;
* have a communicable disease;
* have a biomechanical prosthetic;
* are females who are pregnant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell E Tyler, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- TCNL, 455 Science Drive, Suite 165, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Neuromodulation Rehabilitation: Balance, posture and gait activities; therapeutic exercise for isolated muscle control; transfer training; and relaxation training using neurostimulation modulation. 2-week in lab intervention training, training at home and periodic return for follow-up testing and instruction on the next phase of the intervention.
  Neuromodulation Rehabilitation: Cranial-nerve non-invasive neuromodulation (CN-NINM) uses sequenced patterns of electrical stimulation on the tongue. The hypothesis is that CN-NINM induces neuroplasticity by noninvasive stimulation of two major cranial nerves: trigeminal, CN-V, and facial, CN-VII.
Period: Overall Study
Arm/Group | Neuromodulation Rehabilitation
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Neuromodulation Rehabilitation: Balance, posture and gait activities; therapeutic exercise for isolated muscle control; transfer training; and relaxation training using neurostimulation modulation. 2-week in lab intervention training, training at home and periodic return for follow-up testing and instruction on the next phase of the intervention.
  Neuromodulation Rehabilitation: CN-NINM uses sequenced patterns of electrical stimulation on the tongue. The hypothesis is that CN-NINM induces neuroplasticity by noninvasive stimulation of two major cranial nerves: trigeminal, CN-V, and facial, CN-VII.
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6
Disease Chronicity [Mean (Standard Deviation); unit: years] | 17.7 (7.4)
EDSS Score [Mean (Standard Deviation); unit: units on a scale] — Participants with MS are assessed by a clinician using the Kurtzke Expanded Disability Status Scale (EDSS). Scores range 0-10 (higher numbers indicate greater disability). Participants scoring 1-4.5 can walk without aid, 5.0-7.0 are walking impaired, scores of 7.5+ indicate wheelchair restriction. EDSS draws on the Kurtzke Functional Systems Scores (FSS) that assess 7 physiologic systems affected by MS. FSS ranges from 0-10 in each subsystem, where higher numbers indicate greater levels of dysfunction. The resulting EDSS characterizes the overall ability of the individual.
  units on a scale | 7.0 (0.4)
MS Subtype [Number; unit: participants] — Secondary Progressing MS (SPMS) follows an initial Relapsing-Remitting (RRMS) diagnosis (~85 percent of initial MS diagnoses), characterized by relapses of increased disease activity and worsening symptoms, followed by remissions when the disease does not progress. SPMS is characterized as a gradual increase in disability as the disease progresses, with or without evidence of relapse or changes in an MRI scan. Primary Progressive MS (PPMS) is occurs in ~15 percent of initial MS diagnoses and presents as a steady progression of the disease with no clear relapses or remissions.
  participants
    SPMS | 5
    PPMS | 1

OUTCOME MEASURES:

1. Primary Outcome: Trunk Impairment Scale (TIS)
Description: Static and dynamic sitting balance and trunk coordination are evaluated by a clinician. It is scored on a scale from 0-23, where the higher the score, the more improved the balance. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, and 21 weeks
Population: Effect sizes from baseline reported for 4 subjects with EDSS 6.5 - 7.0. It was postulated that the physical limitations of two subjects with EDSS score of 7.5 presented special challenges to measuring changes in function with the available assessment mechanisms for this clinical population.
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 0.82
  Baseline to Week 6 | 2.58
  Baseline to Week 11 | 1.47
  Baseline to Week 16 | 1.63
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 3.06

2. Secondary Outcome: Static Standing Balance Test
Description: Clinician measures standing balance for up to 30 seconds in each of 5 conditions: feet 10 cm apart, feet together, stride stance, tandem stance, and single leg stance with eyes open and eyes closed. Total score is the sum of all 5 conditions. Higher scores indicate better balance. Performance-based and tested in participants who possessed the ability to perform the assessment. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 0.90
  Baseline to Week 6 | 0.57
  Baseline to Week 11 | 1.04
  Baseline to Week 16 | 0.90
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 0.49
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | 0.32

3. Secondary Outcome: Impact of Visual Impairment Scale (IVIS)
Description: A 5-item self-report questionnaire that assesses the extent to which various activities dependent upon vision are affected by MS-related visual problems. Scores range from 0-15, with higher scores indicating a greater impact of visual problems on daily activities. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, and 21 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 1.27
  Baseline to Week 6 | 2.12
  Baseline to Week 11 | 3.54
  Baseline to Week 16 | 3.54
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 2.12

4. Secondary Outcome: Medical Outcomes Study (MOS) Pain Effects Scale (PES)
Description: A self-report scale that assesses the ways in which pain and unpleasant sensation interfere with mood, ability to walk or move, sleep, work, recreation, and enjoyment of life. This assessment is used for subjects who have pain. Scores can range from 6-30. Items are scaled so that higher scores indicate a greater impact of pain on a patient's mood and behavior. Symptom specific test, only used for participants who presented symptom. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, and 21 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 0.55
  Baseline to Week 6 | 0.64
  Baseline to Week 11 | 0.71
  Baseline to Week 16 | 0.40
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 1.00

5. Secondary Outcome: Bladder Control Scale (BLCS)
Description: A 4-item self-report scale to evaluate the impact of bladder control on lifestyle. This assessment is used for subjects with bladder issues. Scores can range from 0-22, with higher scores indicating greater bladder control problems. Symptom specific test, only used for participants who presented symptom. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 0.30
  Baseline to Week 6 | 0.30
  Baseline to Week 11 | 0.13
  Baseline to Week 16 | 0.41
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 0.62
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | 0.27

6. Secondary Outcome: Bowel Control Scale (BWCS)
Description: A 5-item self-report scale to evaluate the impact of bowel control on lifestyle. This assessment is used for subjects with bowel issues. Scores can range from 0-26, with higher scores indicating greater bowel control problems. Symptom specific test, only used for participants who presented symptom. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 1.20
  Baseline to Week 6 | 0.68
  Baseline to Week 11 | 0.52
  Baseline to Week 16 | 1.04
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 0.86
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | 0.35

7. Secondary Outcome: Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Description: A brief, clinician-administered test that helps determine the neuropsychological status of adults who have neurologic injury or disease such as dementia, head injury, and stroke. This tool consists of a battery of tests. Raw scores are transformed to a 0-120 scale, with a higher score indicating higher function. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | -0.12
  Baseline to Week 6 | 0.39
  Baseline to Week 11 | 0.24
  Baseline to Week 16 | 0.78
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 1.94
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | 0.51

8. Secondary Outcome: Walking Distance
Description: Clinician measures how far the individual can walk until fatigue requires him/her to stop. Longer distances demonstrate improvement. Performance-based and tested in participants who possessed the ability to perform the assessment. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 0.89
  Baseline to Week 6 | 0.75
  Baseline to Week 11 | 0.76
  Baseline to Week 16 | 0.69
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 0.67
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | 0.26

9. Secondary Outcome: Walking Speed
Description: Assessed by timing the first 25 feet that the person walked. Performance-based and tested in participants who possessed the ability to perform the assessment. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 0.77
  Baseline to Week 6 | 0.84
  Baseline to Week 11 | 1.00
  Baseline to Week 16 | 1.01
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | -0.41
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | -0.94

10. Secondary Outcome: 12-item MS Walking Scale (MSWS-12)
Description: A 12-item self-report measure of the impact of MS on a person's walking. Raw scores are transformed to a 0-100 scale. A reduction in score indicates improvement. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | -0.50
  Baseline to Week 6 | 0.43
  Baseline to Week 11 | 0.87
  Baseline to Week 16 | 0.50
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 1.33
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | -0.42

11. Secondary Outcome: Box & Blocks (B&B) Assessment - Right
Description: A standardized clinical assessment of gross upper limb dexterity. Subjects move small blocks from one side of a box to the other within a time period (one minute). Each side is tested separately. The score is the number of blocks moved from 0-150. A higher score indicates improvement. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 0.52
  Baseline to Week 6 | 0.45
  Baseline to Week 11 | 0.47
  Baseline to Week 16 | 1.17
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 0.21
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | 4.95

12. Secondary Outcome: Box & Blocks (B&B) Assessment - Left
Description: as for outcome 11
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 0.07
  Baseline to Week 6 | 0.50
  Baseline to Week 11 | 0.80
  Baseline to Week 16 | 0.58
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | -0.04
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | 0.00

13. Secondary Outcome: Multiple Sclerosis Impact Scale (MSIS-29) - Physical
Description: A 29-item self-report tool that measures the impact of MS on day-to-day life. There are 3 scores, physical, psychological, and total score. Raw scores are transformed to a 0-100 scale. A higher score indicates a greater impact of disease on daily function. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 1.58
  Baseline to Week 6 | 0.61
  Baseline to Week 11 | 0.94
  Baseline to Week 16 | 0.89
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 1.46
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | -0.71

14. Secondary Outcome: Multiple Sclerosis Impact Scale (MSIS-29) - Psychological
Description: as for outcome 13
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 1.77
  Baseline to Week 6 | 1.17
  Baseline to Week 11 | 0.86
  Baseline to Week 16 | 0.98
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 2.05
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | 0.35

15. Secondary Outcome: Modified Fatigue Impact Scale (MFIS)
Description: A self-report tool that assesses the perceived impact of fatigue on daily activities. Consists of 21 items selected from the Fatigue Impact Scale. Scored on a 0-84 scale. A higher score indicates a greater impact of fatigue on daily activities. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 0.87
  Baseline to Week 6 | 3.10
  Baseline to Week 11 | 2.54
  Baseline to Week 16 | 1.75
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 1.40
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | 0.20

16. Secondary Outcome: Gross Motor Function Measure (GMFM)
Description: The GMFM a standardized observational instrument that measures change in gross motor function. Subscales include lying & rolling; sitting; crawling & kneeling; standing; and walking, running & jumping. For the complete test, the raw scores are converted to a 0-100 scale, with higher scores indicating greater functional mobility. The items that we used were scored on a 0-3 scale and changes reported in percent improvement. Performance-based and tested in participants who possessed the ability to perform the assessment. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 6 | 0.82
  Baseline to Week 11 | 1.10
  Baseline to Week 16 | 1.19
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 0.84
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | 0.16

17. Secondary Outcome: Slump Test
Description: Measures and quantifies changes in trunk control during functional sitting. It was quickly determined that this test duplicated the TIS and was difficult to score objectively so the decision was made not to use it for the study. Performance-based and tested in participants who possessed the ability to perform the assessment.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: The Slump Test was ultimately not used because the investigators decided to use the TIS instead. The TIS was realized to be the more appropriate assessment of the two, and the investigators wanted to avoid both data redundancy and test fatigue
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 0

18. Secondary Outcome: Modified Rivermead Mobility Index
Description: An 8 item assessment that quantifies the ability to perform transfers. It has been validated in persons with stroke and a mixed neurologic population (43% MS). Score is a 0-40 scale. A higher score indicates higher function. Performance-based and tested in participants who possessed the ability to perform the assessment. Effect size is reported (quantified difference between baseline and time point). The larger the absolute value, the stronger the effect. Cohen's guidelines for social sciences indicate 0.10 as a "small" effect size, 0.30 as a "medium" effect size, and 0.50 as a "large" effect size.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of change
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 4
percentage of change
  Baseline to Week 2 | 1.01
  Baseline to Week 6 | 1.21
  Baseline to Week 11 | 0.94
  Baseline to Week 16 | 1.44
  Baseline to Week 21: number analyzed (Participants) | 3
  Baseline to Week 21 | 1.15
  Baseline to Week 27: number analyzed (Participants) | 2
  Baseline to Week 27 | 0.38

19. Other Pre Specified Outcome: Video Nystagmography (VNG)
Description: VNG is a standardized eye tracking test used to measure static and dynamic eye movement control to detect oculomotor abnormalities typically associated with degenerative neurological disorders, particularly in the brainstem and cerebellum. The subject wears goggles while an infrared video camera monitors and records eye movement as the eyes follow a dot on a computer screen.
Time Frame: Change from Baseline at 2, 6, 11, 16, 21 and 27 weeks
Population: The VNG was exploratory and opportunistic. The results are not available as the software to perform the quantitative data analysis is still under development.
Arm/Group | Neuromodulation Rehabilitation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Neuromodulation Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuromodulation Rehabilitation (N=6)
Injury (Injury, poisoning and procedural complications) | 1 (1) — Superficial abrasion on both her right forearm during a follow-up visit to the lab.
Trigeminal Neuralgia (TN) (Nervous system disorders) | 1 (1) — The subject reported that the stimulation seemed to ease the symptoms of TN when she resumed training
Viral Infection (Infections and infestations) | 2 (2)
Fatigue (General disorders) | 1 (1)
Osteoarthritis Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes